CLINICAL TRIAL: NCT04819542
Title: Use of Compression Bandages in the Prevention of Post-mastectomy Lymphoceles
Acronym: BANDOCELE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0350
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Lymphocele
Keywords: mastectomy
MeSH Terms: conditions — Lymphocele | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- drain + compression bandage (Experimental)
  Interventions: Device: Bandage
- drain without compression bandage (Active Comparator)
  Interventions: Device: No bandage

INTERVENTIONS:
Device: Bandage — Bandage
  Arms: drain + compression bandage
Device: No bandage — No bandage
  Arms: drain without compression bandage

SUMMARY:
Lymphocele secondary to a mastectomy whether or not associated with a lymph node procedure (sentinel lymph node or axillary dissection) is an almost systematic consequence observed in the postoperative situation in this type of surgery.

This can be the source of pain, skin complications, and infection with a significant impact on the length of hospitalization for patients treated for breast cancer.

There is no consensus regarding the management of lymphocele. The placement of a compression bandage after mastectomy and / or axillary dissection would allow a more efficient and rapid reduction of the lymphocele and a reduction in recurrences.

This would make it possible to reduce the duration of the wearing of the drain, which determines the length of hospitalization and reduce the recurrence of lymphoceles, the punctures of which can be one of the risk factors for secondary lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old,
* Undergoing mastectomy-type surgery with or without axillary dissection for breast cancer
* Affiliated with a health insurance plan

Exclusion Criteria:

* Recurrence of breast cancer,
* Mastectomy with RMI (immediate breast reconstruction) at the same time of operation
* Anticoagulant treatment at curative dose
* Arteritis obliterans of the upper limbs,
* Other cancer during treatment,
* Decompensated heart failure,
* Acute infectious episode (cellulitis, erysipelas, lymphangitis)
* Acute deep vein thrombosis upper limb ipsilateral to mastectomy,
* Cutaneous atrophy of the upper limb,
* Bullous dermatoses,
* Hyperalgesia of the shoulder
* Inability to submit to the constraints of the protocol,
* Impossibility for the patient to achieve self-restraint at the thoracic level
* Pregnancy,
* Feeding with milk
* BMI> 35
* Adult protected by law (guardianship, curatorship and safeguard of justice).
* Anyone who is not in a position to give their consent in writing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion in percentage of patients treated successfully | 6 months
  Provide an estimate of the proportion of patients treated successfully (success rate defined by the absence of lymphocele on D4 post mastectomy) in two groups of patients (drain + compression bandage vs drain without compression bandage).

SECONDARY OUTCOMES:
Lymphocele volume in milliliter | 6 months
  Lymphocele volume at day 4, day 8 and 6 months post mastectomy
Number of lymphocele punctures | 6 months
  Number of lymphocele punctures possibly performed during the 6 months of follow-up
Clinical signs associated with lymphocele | 8 days
  Clinical signs associated with lymphocele at day 4 and day 8 (redness, blister, local inflammation (erythema + redness + warmth), rash, pruritus, ecchymosis, wound, allergic reaction, presence of clinical lymphocele, pain in the limb ipsilateral on surgery, heaviness in the ipsilateral limb discomfort when using the ipsilateral limb, perimeter measurements (in centimeters) at the level of both upper limbs using a standard seamstress ruler, measurement of joint amplitudes (in centimeters).
Frequency of adverse events | 6 months
  The frequency of adverse events during the 6-month follow-up
Clinical signs associated with lymphocele | 8 days
  Clinical signs associated with lymphocele at day 4 and day 8 : perimeter measurements (in centimeters) at the level of both upper limbs using a standard seamstress ruler
Clinical signs associated with lymphocele | 8 days
  Clinical signs associated with lymphocele at day 4 and day 8 : measurement of joint amplitudes (in centimeters).
Changes in quality of life | 6 months
  Changes in quality of life, with QLQ-C30 questionnaire, (specifically linked to breast cancer and overall quality of life) at day 8, day 21 and at 6 months post mastectomy, compared to an assessment before mastectomy
Changes in quality of life | 6 months
  Changes in quality of life, with 5Q-5D-5L questionnaire, (specifically linked to breast cancer and overall quality of life) at day 8, day 21 and at 6 months post mastectomy, compared to an assessment before mastectomy

CONTACTS AND LOCATIONS:
Overall Officials: Julie MALLOIZEL DELAUNAY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No